CLINICAL TRIAL: NCT04818788
Title: Hematological Indices and Fecal Calprotectin as Predictors of Histological Remission in Ulcerative Colitis Patients Receiving Biological Therapy
Brief Title: Hematological Indices and Fecal Calprotectin Predict Histological Remission in Ulcerative Colitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdallah Abdelfadil Abdelal, internal medicine physician, Assiut University
Other Study IDs: ulcerative colitis
Record Dates: First submitted 2021-03-20; First posted 2021-03-26 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Biological Drug — we will give biological drugs to indicated ulcerative colitis patients and we will investigate the predictive ability of fecal calprotectin and hematological indices to histological remission

SUMMARY:
Investigators aimed at investigating the prediction ability of faecal calprotectin to predict mucosal healing and histological remission in ulcerative colitis patients receiving biological therapy Investigators aimed to evaluate the prediction ability of NLR, PLR and MLR to predict mucosal healing and histological remission in ulcerative colitis patients receiving biological therapy.

Investigators evaluate the histological remission in ulcerative colitis patients receiving biological therapy in Assuit university hospital.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic relapsing disease that involves the colorectal mucosa. Over the years, the therapeutic target has been upgraded from the resolution of symptoms to deep remission to prevent relapses and complications. The primary therapeutic target to be achieved in patients with UC is both clinical and endoscopic remission . The assessment of histological inflammation has emerged as a promising endpoint in UC . However, the link between histological disease activity and other measures of clinical disease activity is not yet well established . Some authors suggest that the presence of histological inflammation is a better predictor of future clinical relapse than endoscopic activity . Several studies showed that patients with residual microscopic active inflammation seem to be more prone to relapse when compared with patients with normal histology .

Calprotectin is a 36-kDa calcium- and zinc-binding protein, which represents approximately 60% of soluble proteins of granulocyte cytoplasm . Fecal calprotectin (FC) is strongly correlated with both MES and Ulcerative Colitis Endoscopic Score (9, 10). In previous studies, FC was shown to be helpful in predicting sustained clinical remission and mucosal healing during anti-TNF treatment, particularly with IFX and ADA. However, no investigations have been performed to evaluate the predictive value of FC in terms of mucosal healing in a prospective cohort of patients with UC treated with biological therapy. Based on the above background, the aim of the present prospective study is to identify a reliable biomarker able to predict therapeutic effectiveness in UC .

Ulcerative colitis (UC) is a chronic relapsing disease characterized by a neutrophil-mediated inflammation of the gut.

Indeed, European Crohn and Colitis Organization guidelines have highlighted how the grade of neutrophilic infiltration is necessary for the diagnosis of this pathological condition and for the evaluation of histological activity. Thus, colonoscopy is necessary to collect mucosal biopsies and assess neutrophilic infiltration for the diagnosis and during follow-up to evaluate treatment response and predict long-term outcome, although histological healing is still debated. However, colonoscopy is an invasive, costly, and not always well-tolerated examination for patients. Apart from endoscopic interventions, disease severity can be also assessed using less-invasive biomarkers, including blood count.

In these regard the investigators aimed to investigate the ability of prediction of hematological indices including (PLR, NLR and MLR) and fecal calprotectin to predict histological remission in ulcerative colitis patients receiving biological therapy .

ELIGIBILITY:
Inclusion Criteria:

* 24 patients (males and females at the age between 18 and 55 years) of ulcerative colitis indicated to biological therapy

Exclusion Criteria:

* - Ulcerative colitis pregnant women
* Patient receiving biological therapy for extra intestinal manifestation
* Patients on corticosteroids more than 20 mg as it affects leucocytic count
* Patients under the age of 18 years

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: our study will include ulcerative colitis patients who are indicated to biological therapy at gastro enterology unit in internal medicine department at Assuit university during the period of April 2021 to April 2022 and we will do the following to every patient :
  full history including drug history full examination colonoscopy and histological examination before the biological therapy and after 8 weeks and after 25 weeks and after 52 weeks ESR , CRP , Fecal calprotectin and CBC including NLR, PLR and MLR before starting biological therapy and after 8 weeks and after 25 weeks and after 52 weeks
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-04-20 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Histological remission in ulcerative colitis patients receiving biological therapy | one year
  Assessment of histological remission by using Geboes score index Histological remission was defined as Geboes index ≤ 3.0.15 .The Geboes index consists of a scoring system with five distinctive grades [each with subgrades], corresponding to different aspects of inflammatory activity in the mucosa. Grade 0 corresponds to structural [architectural] change, grade 1 to chronic inflammatory infiltrate, grade 2 to lamina propria eosinophils [2A] and neutrophils [2B], grade 3 to neutrophils in the epithelium, grade 4 to crypt destruction, and grade 5 to erosion or ulceration. Higher subgrade scores reflect a more severe condition.
Assessment of fecal calprotectin level in ulcerative colitis patients receiving biological therapy | one year
  measured by quantative enzyme immuno assay μg/g.
Assessment of the level of PLR, NLR , MLR in ulcerative colitis patients receiving biological therapy | one year
  by extraction of the values of blood counts in particular WBC and platelet count
Ability of hematological indices and fecal calprotectin to predict histological remission | one year
  by correlate the level of hematological indices and fecal cal peotectin with histological remission

REFERENCES:
- [Background] Bertani L, Rossari F, Barberio B, Demarzo MG, Tapete G, Albano E, Baiano Svizzero G, Ceccarelli L, Mumolo MG, Brombin C, de Bortoli N, Bellini M, Marchi S, Bodini G, Savarino E, Costa F. Novel Prognostic Biomarkers of Mucosal Healing in Ulcerative Colitis Patients Treated With Anti-TNF: Neutrophil-to-Lymphocyte Ratio and Platelet-to-Lymphocyte Ratio. Inflamm Bowel Dis. 2020 Sep 18;26(10):1579-1587. doi: 10.1093/ibd/izaa062. PMID 32232392
- [Background] Magro F, Lopes SI, Lopes J, Portela F, Cotter J, Lopes S, Moreira MJ, Lago P, Peixe P, Albuquerque A, Rodrigues S, Silva MR, Monteiro P, Lopes C, Monteiro L, Macedo G, Veloso L, Camila C, Afonso J, Geboes K, Carneiro F; Portuguese IBD group [GEDII]. Histological Outcomes and Predictive Value of Faecal Markers in Moderately to Severely Active Ulcerative Colitis Patients Receiving Infliximab. J Crohns Colitis. 2016 Dec;10(12):1407-1416. doi: 10.1093/ecco-jcc/jjw112. Epub 2016 May 25. PMID 27226417
- [Background] Bertani L, Blandizzi C, Mumolo MG, Ceccarelli L, Albano E, Tapete G, Baiano Svizzero G, Zanzi F, Coppini F, de Bortoli N, Bellini M, Morganti R, Marchi S, Costa F. Fecal Calprotectin Predicts Mucosal Healing in Patients With Ulcerative Colitis Treated With Biological Therapies: A Prospective Study. Clin Transl Gastroenterol. 2020 May;11(5):e00174. doi: 10.14309/ctg.0000000000000174. PMID 32677804
- [Background] Okba AM, Amin MM, Abdelmoaty AS, Ebada HE, Kamel AH, Allam AS, Sobhy OM. Neutrophil/lymphocyte ratio and lymphocyte/monocyte ratio in ulcerative colitis as non-invasive biomarkers of disease activity and severity. Auto Immun Highlights. 2019 May 15;10(1):4. doi: 10.1186/s13317-019-0114-8. eCollection 2019 Dec. PMID 32257060